CLINICAL TRIAL: NCT02995291
Title: Reversing the Effects of 0.5% Bupivacaine: A Randomized Controlled Trial
Brief Title: Reversing the Effects of 0.5% Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Pierre-Luc Michaud, Assistant Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-4014
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Phentolamine; Saline Waters

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): 1.7ml saline water
  Interventions: Drug: Saline Water (Control)
- OraVerse (Experimental): 1.7ml OraVerse
  Interventions: Drug: OraVerse

INTERVENTIONS:
Drug: OraVerse — 1.7ml OraVerse (0.4 mg phentolamine mesylate) will be injected once after the participants are found to be well anesthetized following an injection of 1.8ml Bupivacaine 0.5% (inferior alveolar nerve block). Oraverse will be injected at the same site Bupivacaine was injected.
  Other Names: phentolamine mesylate
  Arms: OraVerse
Drug: Saline Water (Control) — 1.7ml saline water will be injected once after the participants are found to be well anesthetized following an injection of 1.8ml Bupivacaine 0.5% (inferior alveolar nerve block). The water will be injected at the same site Bupivacaine was injected.
  Other Names: Placebo
  Arms: Control

SUMMARY:
Clinical trials have shown phentolamine mesylate (PM), brand name OraVerse, to be effective at reducing the amount of time to reversal of local anesthesia with different dental anesthetics. However, to date no study investigated the efficacy of phentolamine mesylate to reverse anesthesia induced with the use of Bupivacaine.

The objective of the proposed research is to conduct a pilot-scale randomized clinical trial evaluating the difference in time required for the return of normal soft-tissue sensation and function in participants who have received 0.5% Bupivacaine HCl, 1:200,000 epinephrine, followed by an injection with either 1) OraVerse (phentolamine mesylate) or 2) sterile physiological water (control).

DETAILED DESCRIPTION:
Dental procedures often require the use of local anesthesia. The most common local anesthetic used is 2% Lidocaine 1:100,000 epinephrine. This local anesthetic can achieve soft tissue anesthesia for 180-300 minutes and pulpal anesthesia for 60 minutes. Unfortunately, for longer treatments this relatively short duration can lead to the loss of anesthetic effect before the end of the interventions. Time-demanding dental appointments include oral and periodontal surgeries, extensive restorative treatments, and even minor treatments when completed by dental students. Unfortunately, if a short acting anesthetic such as Lidocaine is being used during long lasting procedures, once the patients start feeling pain again, it may be difficult to reestablish deep pulpal anesthesia with a repeated injection due to tachyphylaxis. To avoid this situation long-acting local anesthetics could be selected instead. The only long-acting anesthetic available in dentistry is 0.5% Bupivacaine HCl, 1:200,000 epinephrine. Bupivacaine can produce soft tissue anesthesia for up to 12 hours (commonly 4 to 9 hours) and pulpal anesthesia for up to 7 hours (commonly 1.5 to 3 hours). Unfortunately, Bupivacaine is not often used for non-surgical procedures due to its very long soft tissue anesthesia that outlast treatments by several hours.

The effects of soft tissue anesthesia linger for some time after the administration of long acting local anesthetics such as Bupivacaine. This can lead to discomfort and occasionally injury from lip/tongue biting. Clinical trials have shown phentolamine mesylate (PM), brand name OraVerse, to be effective at reducing the amount of time to reversal of local anesthesia with different dental anesthetics. However, to date no study investigated the efficacy of phentolamine mesylate to reverse anesthesia induced with the use of Bupivacaine.

The objective of the proposed research is to conduct a pilot-scale randomized clinical trial evaluating the difference in time required for the return of normal soft-tissue sensation and function in participants who have received 0.5% Bupivacaine HCl, 1:200,000 epinephrine, followed by an injection with either 1) OraVerse (phentolamine mesylate) or 2) sterile physiological water (control). This will further advance our knowledge of both Bupivacaine and phentolamine mesylate as there are no current studies evaluating reversing the effect of Bupivacaine with PM.

It is hypothesized that phentolamine mesylate will reduce the duration of soft tissue anesthesia by 2.5 hours when compared with a control injection of saline water. It is anticipated that this study will determine the feasibility and sample size needed to conduct a full-scale multi-centre trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* capable of providing informed consent

Exclusion Criteria:

* contra-indications for regular dental treatment
* medical history that contraindicates the use of epinephrine
* participant taken an opioid or an opioid like analgesic within 24 hours
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Time to reversal of local anesthesia | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Luc Michaud, DMD, MSc, FRCDC, Principal Investigator — Dalhousie University
Locations (1):
- Dalhousie University Faculty of Dentistry, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate data to be published in peer reviewed journal

REFERENCES:
- See also: Dalhousie University Faculty of Dentistry Web Site — http://www.dal.ca/faculty/dentistry.html